CLINICAL TRIAL: NCT00942838
Title: Whole Abdomen Radiation in Conjunction With Intraperitoneal Chemotherapy for the Treatment of Small Volume Recurrent Ovarian Carcinoma Limited to the Peritoneal Cavity: A Phase I Trial
Brief Title: Whole Abdomen Radiation in Conjunction With Intraperitoneal Chemotherapy for the Treatment of Small Volume Recurrent Ovarian Carcinoma Limited to the Peritoneal Cavity
Acronym: WAR
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decision due to under accrual.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI28777
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Recurrent Ovarian Carcinoma
Keywords: Recurrent Ovarian Carcinoma; Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cisplatin — PLATINOL®-AQ (cisplatin injection) is a clear, colorless, sterile aqueous solution, each mL containing 1 mg cisplatin and 9 mg Sodium Chloride, USP. HCl and/or Sodium Hydroxide is added to adjust pH of the solution. The active ingredient, cisplatin, is a yellow to orange crystalline powder with the molecular formula PtCl2H6N2, and a molecular weight of 300.1. Cisplatin is a heavy metal complex containing a central atom of platinum surrounded by two chloride atoms and two ammonia molecules in the cis position. It is soluble in water or saline at 1 mg/mL and in dimethylformamide at 24 mg/mL. It has a melting point of 207°C.
  Other Names: Cisplatin, PLATINOL®-AQ
Radiation: Whole Abdomen Radiotherapy — Whole abdominal radiotherapy will be delivered with an open-field anterior-posterior/posterior-anterior technique. Radiation will be administered in a dose escalating fashion to determine toxicity. The maximal dose of radiation will be defined as a mean midplane dose to the abdomen of 3,000 Gy through parallel-opposed single ports with a 1-cm margin that will cover the entire abdomen including the diaphragm.
  Other Names: radiation therapy

SUMMARY:
The proposed study is a prospective cohort study incorporating patients with first recurrence ovarian or primary peritoneal cancer who will receive intraperitoneal chemotherapy in conjunction with whole abdomen radiation. The primary end point of this investigator initiated research study is to determine the toxicity associated with whole abdomen radiation in combination with intraperitoneal chemotherapy.

Primary Objective:

* Determine the maximum tolerated dose (MTD) of whole abdomen radiation in conjunction with intraperitoneal cisplatin chemotherapy in the treatment of women with small volume (< 1 cm) recurrent ovarian cancer confined to the abdominal peritoneal cavity.

Secondary Objective:

* Quality of Life assessment.

DETAILED DESCRIPTION:
DESIGN: This is an open label, single arm, dose finding study.

STUDY PROCEDURES: Patients will receive chemotherapy and radiation for four weeks, and we will check for any problems from the treatment for 3 months. We would like to collect information from the patients regular doctor for 1 year after this treatment.

Pre-screening If patients decide to participate in this study the doctor will evaluate if they have met all the criteria to be eligible. To participate the cancer cannot have spread outside the abdomen and patients must have had only one type of chemotherapy for their cancer. If there any of their previous scans or blood tests show that the cancer has spread outside the abdominal cavity, patients will not be able to participate in this study. Patients will also not be able to participate in this study if it is determined that their cancer has come back less than six months after they completed their first treatment of chemotherapy. If these criteria are met, the standard next step for treatment is to have a second surgery to remove all or most of the cancer from the abdominal cavity. This will involve a similar surgery to what patients had when their cancer was first diagnosed. During this surgery we will place a special catheter or tube within the abdominal cavity so that we can administer chemotherapy into the abdomen directly and deliver it to the remaining cancer.

Screening Procedures:

The following screening tests, exams and procedures will be done:

* Recording of medical history, physical exam (including vital signs, height & weight assessment, pelvic examination)
* Blood tests (approximately 2-3 teaspoons will be drawn)
* Urine tests
* Quality of life questionnaire
* If patients have a history of hearing loss, they will have a hearing test because cisplatin can affect hearing.

Chemotherapy and Radiation Treatment:

* Chemotherapy (Cisplatin) will be given to after recovery from surgery. It will be given once per week at the same time as patients begin receiving the radiation treatment for the first 4 weeks. The chemotherapy will be given through the catheter (tube) that was placed under the skin during surgery and will not be visible. Patients will receive medication prior to the chemotherapy to prevent nausea, vomiting, and possible allergic reaction. Each infusion of chemotherapy will take approximately 60 minutes. After patients receive the drug we will ask to change positions to ensure that the drug comes in contact with all parts of the abdomen.
* Radiation therapy will be administered for four weeks. Radiation treatments will be given every day (Monday through Friday) for approximately four weeks.
* Weekly blood tests will be taken before patients receive the chemotherapy (approximately 2-3 teaspoons) to monitor the effects of the drug on the body.
* The study doctor will evaluate patients weekly with a physical exam and review their blood tests for any side effects they might be having from the chemotherapy or radiation treatments.
* Complete a quality of life questionnaire each week.

At the end of treatment (beginning of week 5) AND approximately 90 days after the completion of treatment patients will have a physical exam, blood tests evaluation of the side effects, and will complete a quality of life questionnaire.

At the end of treatment, patients will likely undergo additional standard chemotherapy treatment. We would like to collect and review the information about their progress and care for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent ovarian cancer or primary peritoneal cancer with disease confined to the abdomen and pelvis, who have undergone optimal cytoreductive surgery for recurrence
2. Must have received only one prior chemotherapeutic regimen as their prior therapy
3. Eligible patients must have received platinum based intravenous chemotherapy as their only prior therapy. Previous treatment with maintenance chemotherapy after initial adjuvant chemotherapy is acceptable, including anti-estrogen therapy and growth factors. Previous intraperitoneal chemotherapy is not allowed
4. Patients have evidence of recurrent cancer manifested by either a) elevation in serum CA-125 or a palpable tumor on physical exam and/or b) radiographic evidence of recurrence. (Note that a tissue biopsy for histologic confirmation of tumor recurrence prior to cytoreductive surgery is not necessary, however histologic confirmation of the removed tumor is necessary- see exclusion 5.22)
5. Tumors with serous, mucinous, clear cell, or endometrioid histologic types are eligible
6. Recurrent disease must be confined to the abdominal cavity
7. Recurrence of tumor must be greater than six months from completion of primary chemotherapy (platinum sensitive ovarian cancer)
8. Patients have undergone a second cytoreductive surgery to remove all gross residual disease. This cytoreductive surgery must occur within twelve weeks of enrollment
9. Patients have or are planning to have an IP catheter
10. Patients who require rectosigmoid resection with primary anastamosis will be eligible
11. Adequate renal function as defined by serum creatinine less 2.0mg/dL
12. Patients must have appropriate hematologic parameters with total white blood cell (WBC) counts ≥ 3,000cells/mcl and platelet counts ≥ 100,000/mcl prior to treatment initiation
13. Patients must have the absence of pleural effusions on chest radiographs
14. Patients must sign informed consent approved by the University of Utah and institutional review board (IRB)
15. ECOG performance status less than or equal to 2
16. Age greater than 18 years old

Exclusion Criteria:

1. Patients previously characterized with stage IV disease or those with stage IIIC who underwent suboptimal secondary cytoreductive surgery for recurrence will not be eligible for participation
2. Patients who undergo secondary cytoreductive surgery for recurrence and have no recurrent disease by histologic documentation will not be eligible
3. Those with preoperative evaluation consistent with stage IV disease (pleural effusion or liver parenchymal disease)
4. Patients with disease outside the peritoneal cavity including disease in the thorax, within the parenchyma of the liver, spleen, or retroperitoneal nodal disease will not be eligible for participation
5. Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy
6. Patients determined to have platinum resistant ovarian or primary peritoneal cancer
7. Those who had suboptimal cytoreductive surgery at the time of first diagnosis. This includes patients who had a suboptimal cytoreductive surgery followed by chemotherapy, then a secondary debulking and now have a recurrence
8. Those with > 1cm residual disease after the second cytoreductive surgery
9. Patients that have been treated with previous intraperitoneal chemotherapy
10. Patients that are pregnant or lactating
11. Patients with peripheral neuropathy greater than grade 2 at baseline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of whole abdomen radiation in conjunction with intraperitoneal cisplatin chemotherapy in the treatment of women with small volume (< 1 cm) recurrent ovarian cancer confined to the abdominal peritoneal cavity | 2 years after study start

SECONDARY OUTCOMES:
Quality of Life assessment | 2 years after study start

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P. Soisson, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States